CLINICAL TRIAL: NCT06558760
Title: Continuous Decline in Open Appendectomies to 0.9% and Conversions to 2%
Brief Title: Changes in the Treatment of Acute Appendicitis
Acronym: TreatApp
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Collaborators: CLINOTEL Hospital Association Germany (Unknown)
Responsible Party: Principal Investigator, Habil Claus Schildberg, Principal investigator, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: TreatApp
Record Dates: First submitted 2024-08-07; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Acute Appendicitis
Keywords: Acute Appendicitis; Type of appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to analyse the epidemiology, diagnostics, the type of surgical techniques and their development over time, and mortality in acute appendicitis in 68 hospitals in Germany based on routine data between 2010 and 2022.

DETAILED DESCRIPTION:
This retrospective observational study analyzed routine data provided by the CLINOTEL Hospital Association Germany, covering the years 2010 to 2022. The data was derived from anonymized billing data according to the German Diagnosis-Related Groups (DRG) system for inpatient hospital treatments.

The study focused on the use of different surgical techniques for appendectomy over time, the in-hospital mortality rates and postoperative complications associated with the performed kind of appendectomy.

Patients over 18 years with an acute appendicitis were included by collecting following data: patient demographic, comorbidity, performed operation, postoperative complications, admission to Intensive Care Unit, length of stay, and in-hospital-mortality. Cases without an appendectomy, with nonspecific appendectomy and those, who underwent appendectomy as part of another surgical procedure, were excluded. Furthermore, all cases with multiple appendectomy codes were removed from the sample. Ultimately, 31988 patients were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Acute Appendicitis

Exclusion Criteria:

* Age under 18 years
* No appendectomy performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute appendicitis in 68 hospitals in Germany collected by routine data between 2010 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 31988 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in surgical techniques over time | 2010-2022
  Development of the use of surgical techniques (open, laparoscopic or conversion from open to laparoscopic)

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not available for data sharing.

REFERENCES:
- [Derived] Schildberg C, Weber U, Konig V, Linnartz M, Heisler S, Hafkesbrink J, Fricke M, Mantke R. Laparoscopic appendectomy as the gold standard: What role remains for open surgery, conversion, and disease severity? : An analysis of 32,000 cases with appendicitis in Germany. World J Emerg Surg. 2025 Jun 18;20(1):53. doi: 10.1186/s13017-025-00626-2. PMID 40533760